CLINICAL TRIAL: NCT05185154
Title: Natural Course and Prognosis of Hospitalized Patients With Cirrhosis: a Prospective, Multicenter, and Observational Study
Brief Title: Natural Course and Prognosis of Hospitalized Patients With Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Won Sohn, Principal Investigator, Kangbuk Samsung Hospital
Other Study IDs: KBSMCLC2021
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective study is to evaluate the natural course and prognosis of hospitalized patients with liver cirrhosis.

DETAILED DESCRIPTION:
The aim of this prospective study is to collect data on hospitalized patients with liver cirrhosis at four institutions in Korea (Kangbuk Samsung Hospital, Hallym University Dongtan Sacred Heart Hospital, Chosun University Hospital, and National Medical Center). If patients agree to participate in this clinical trial, the patients' data (such as age, sex, height, weight, nutrition status [RFH-NPT], history of medication, laboratory findings, endoscopic findings, and radiologic findings) will be collected in a research database. The research database will be updated, every 6 months, to include data on patients' disease outcomes and follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with liver cirrhosis
* Admission to the hospital because of cirrhotic complications such as uncontrolled ascites, variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, spontaneous bacterial peritonitis, hepatocellular carcinoma, acute kidney injury, bacterial infection, acute liver failure, and etc.

Exclusion Criteria:

* Admission to the hospital without cirrhotic complications
* Patients who refuse the follow-up of outpatient department

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with liver cirrhosis
Sampling Method: Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Up to 2 years
  Death from any cause
Liver-related mortality | Up to 2 years
  Death from liver disease

SECONDARY OUTCOMES:
Cause of admission to hospital | At baseline
  Prevalence of cause of admission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Won Sohn, MD, PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (4):
- South Korea (4):
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Chosun University Hospital, Kwangju
  - Jae Yoon Jeong, Seoul
  - Kangbuk Samsung Hospital, Seoul